CLINICAL TRIAL: NCT06414304
Title: A Multi-center Observational Clinical Trial Evaluating the Dynamics of Microsatellite Instability and Genomic Profile of Colorectal Cancer in the Course of Treatment With Immune Checkpoint Inhibitors
Brief Title: Dynamics of MSI and Genomic Profile of Colorectal Cancer In the Course of Immune Checkpoint Inhibitor Therapy
Acronym: BLOOMSI
Status: Completed | Type: Observational
Sponsor: OncoAtlas LLC (Industry)
Collaborators: N.N. Blokhin National Medical Research Center of Oncology (Other); Moscow MultidisciplinaryClinical Center Kommunarka (Unknown)
Responsible Party: Sponsor
Other Study IDs: BLOOMSI; 22-75-10154 (Other Grant/Funding Number: Russian Science Foundation)
Record Dates: First submitted 2024-05-07; First posted 2024-05-16 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Colorectal Cancer; Colorectal Cancer Metastatic; MSI-H Colorectal Cancer; dMMR Colorectal Cancer; Cancer; Colon Adenocarcinoma
Keywords: MSI; dMMR; Microsatellite instability; Next-generation sequencing; Immunotherapy; Immune checkpoint inhibitors; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Colonic Neoplasms; Microsatellite Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
Colorectal cancer (CRC) is a leading cause of cancer-related mortality worldwide. Microsatellite instability or mismatch repair deficiency occurs in 20% of CRC, and is predominantly found in non-metastatic tumors. The success of the CheckMate 142 and KEYNOTE-177 clinical trials has shifted the treatment paradigm of the MSI/dMMR CRC, which has led to the adoption of immune checkpoint inhibitors (ICI) by international treatment standards. However, despite the encouraging effects of ICI, up to 30% of patients are resistant to treatment and exhibit rapid disease progression shortly after starting ICI. On the other hand, around 30% of patients treated with ICI demonstrate prolonged responses to the treatment with a duration of response of over 40 months. Furthermore, for ~10% of patients, treatment with ICI results in pseudo-progression - a phenomenon of a short-term increase followed by the decrease of the tumor volume.

Currently, the mechanisms and biomarkers associated with the response or resistance to ICI in MSI-positive CRC are largely unknown. Select studies suggest that BRAF mutations (specifically, BRAF p.V600E) might negatively affect the patients' progression-free survival following ICI, however, these data are premature.

The primary hypothesis is that the clonal heterogeneity and the evolution of MSI status of MSI-positive CRC will play a role in the development of ICI treatment resistance. The primary objective of the study is to investigate the dynamics of MSI status in serial liquid biopsy samples from patients with MSI-positive tumors receiving ICI.

DETAILED DESCRIPTION:
This is a multicenter observational trial designed to evaluate the dynamics of microsatellite instability and the genomic profiles of CRC during immune checkpoint inhibitor treatment.

Patients with MSI/dMMR-positive tumors who are candidates for the ICI treatment will be included in the study. MSI/dMMR positivity should be confirmed with polymerase chain reaction-based (PCR) assays, immunohistochemistry (IHC) or Next-generation sequencing (NGS). Treatment with any ICI will be allowed. Upon inclusion in the study, patients will be asked to provide the pre-treatment FFPE tumor and liquid biopsy (LB) samples along with LB samples on the 14th, 28th days of ICI, and at every control study. LB samples will be collected until treatment discontinuation.

The pre-treatment FFPE samples will be tested with an alternative routine method (PCR and/or IHC, depending on what method was used for initial testing), as well as with the Solo Atlas Pro NGS panel covering common cancer-related genes and short tandem repeats for MSI detection. All LB samples will be tested with the Solo Atlas Pro NGS panel. Dynamics of MSI and genomic profiles will be correlated with the treatment outcomes.

Disease response to study treatment will be evaluated by imaging methods. Response to treatment will be determined by RECIST v1.1.

ELIGIBILITY:
Inclusion Criteria:

* Male/female participants must be at least 18 years of age on the day of signing informed consent and have a histologically confirmed diagnosis of colorectal cancer.
* Verified MSI/dMMR positivity as measured by 5-loci PCR or 4-antibody IHC.
* The patient is scheduled to start treatment with any of the immune checkpoint inhibitors 2-4 weeks after the inclusion in the study.
* Have provided an archival tumor tissue sample obtained prior to the start of treatment with immune checkpoint inhibitor(s). Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides.
* Patient has to be able to provide serial blood samples during the course of treatment, as well as on every follow-up tumor scan.
* The participant (or legally acceptable representative if applicable) provides written informed consent to participate in the trial.
* Have measurable disease based on RECIST 1.1.
* Have adequate organ function.

Exclusion Criteria:

* Prior treatment with immune checkpoint inhibitors.
* For female participants: pregnancy or planned pregnancy.
* The unavailability of the tumor or serial liquid biopsy samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed colorectal cancer with microsatellite instability (MSI) or mismatch repair deficiency (dMMR)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Concordance of NGS and routine methods (PCR, IHC) for MSI analysis | Through study completion, an average of 3 years
  Concordance will be calculated using Cohen's Kappa (κ)

SECONDARY OUTCOMES:
Concordance of MSI in tumor tissue and liquid biopsy (ctDNA) | Through study completion, an average of 3 years
  Concordance will be calculated using Cohen's Kappa (κ)
Qualitative and quantitative status of MSI in serial liquid biopsy (ctDNA) samples | Through study completion, an average of 3 years
  Liquid biopsy samples will be collected prior to the start of ICI, on the 14th and 28th days of therapy and at every follow-up tumor scan

OTHER OUTCOMES:
Correlation of biomarkers with the treatment outcomes | Through study completion, an average of 3 years
  Dynamics of biomarkers in serial liquid biopsy samples will be correlated with treatment outcomes. Response to treatment will be determined by RECIST v1.1.
Evaluation of the ctDNA dynamics in the course of ICI in serial plasma samples | Through study completion, an average of 3 years
  Dynamics of ctDNA in serial liquid biopsy samples will be correlated with treatment outcomes. Response to treatment will be determined by RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Ivanov, PhD, Principal Investigator — OncoAtlas LLC
Locations (2):
- Russia (2):
  - N.N.Blokhin National Medical Research Center of Oncology, Moscow
  - State Budgetary Institution of Healthcare of the City of Moscow "Moscow Multidisciplinary Clinical Center "Kommunarka" of the Department of Health of the City of Moscow, Moscow